CLINICAL TRIAL: NCT05329597
Title: Study on Pharmacokinetics and Gene Polymorphism of Umorestat Hydrogen Sulfate Capsule in Patients With Locally Advanced/Metastatic Pancreatic Cancer
Brief Title: Study on Umorestat Hydrogen Sulfate Capsule in Patients With Locally Advanced/Metastatic Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: 2020-KY-040
Record Dates: First submitted 2021-12-21; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Pharmacokinetics; Pancreatic Cancer; Gene Polymorphisms
Keywords: pharmacokinetics; gene polymorphisms; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This experiment involves genotyping of blood cells。
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 100mg: After 15 consecutive days of takeing 100mg Umorestat capsule of each participant, 2 mL of peripheral venous blood is collected at 3 h, 8 h and 24 h (D16) on the 15th day into the vacuum blood collection tube via EDTA anticoagulation for genotyping and metabolite determination.
  Interventions: Genetic: Genotyping
- 200mg: After 15 consecutive days of takeing 200mg Umorestat capsule of each participant, 2 mL of peripheral venous blood is collected at 3 h, 8 h and 24 h (D16) on the 15th day into the vacuum blood collection tube via EDTA anticoagulation for genotyping and metabolite determination.
  Interventions: Genetic: Genotyping
- 400mg: After 15 consecutive days of takeing 400mg Umorestat capsule of each participant, 2 mL of peripheral venous blood is collected at 3 h, 8 h and 24 h (D16) on the 15th day into the vacuum blood collection tube via EDTA anticoagulation for genotyping and metabolite determination.
  Interventions: Genetic: Genotyping
- 600mg: After 15 consecutive days of takeing 600mg Umorestat capsule of each participant, 2 mL of peripheral venous blood is collected at 3 h, 8 h and 24 h (D16) on the 15th day into the vacuum blood collection tube via EDTA anticoagulation for genotyping and metabolite determination.
  Interventions: Genetic: Genotyping

INTERVENTIONS:
Genetic: Genotyping — Genotyping is performed using the subjects' blood cells

SUMMARY:
Based on the tolerability, safety and pharmacokinetics phase I/II clinical trials of ulimostat hydrochloride capsules (LH011) combined with gemcitabine hydrochloride (GEM) in locally advanced/metastatic pancreatic cancer patients, to determine pharmacokinetics, the biotransformation pathway and metabolite profile of ulimostat in patients with locally advanced/metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This study is a research on the pharmacokinetics and gene polymorphisms of ulimostat hydrochloride capsules in patients with locally advanced/metastatic pancreatic cancer. Aims to collect the "Phase I/II clinical trials of the tolerability, safety and pharmacokinetics of ulimostat capsules (LH011) combined with gemcitabine hydrochloride (GEM) in patients with locally advanced/metastatic pancreatic cancer" patient's peripheral blood sample to determine the structure of the metabolites of ulimostat in the biological samples and trough concentration and genotyping tests were performed on patients to investigate the correlation between gene polymorphisms of metabolic enzymes, transporters, target protein uPA and proteins expressed in upstream and downstream signaling pathways and blood drug concentration, efficacy, safety and tolerance of ulimostat.

ELIGIBILITY:
Inclusion Criteria:

* Successfully enrolled in a Phase I/II clinical study on the tolerability, safety and pharmacokinetics of Umorestat hydrogen Sulfate capsule (LH011) combined with gemcitabine hydrochloride (GEM) for patients with locally advanced/metastatic pancreatic cancer.
* Fully understand the purpose and requirements of this study and sign a written informed consent.
* Willing to provide blood samples.

Exclusion Criteria:

* Suffering from inflammatory bowel disease.
* The researcher considers it unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients With Locally Advanced/Metastatic Pancreatic Cancer
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Metabolite profile | After sampling blood samples (approximately 2 weeks)
  Determine the drug metabolite profile: Serum samples were detected by ultra-high pergormance liquid tandem chromatography quadrupole time of flight mass spectrometry(LC-MS). Differential metabolites were screened by principal component analysis(PCA), orthogonal projections to latent structures-discriminant analysis(OPLS-DA) and Student's t-test. Then the hierarchical clustering analysis(HCA) was carried out for the screened differential metabolites.
Genotyping | After sampling blood samples (approximately 2 weeks)
  To determine the relationship between genotyping and drug exposure, efficacy and safety: Employs PCR to amplify the regions of the genome containing each SNP, then use MassARRAY to detect mass differences between fragments differing by a single base. Use genotyping test results to do correlation analysis with drug concentration, safety results, and efficacy results to determine the relationship between different types of gene locus mutations and drug concentration, efficacy, and adverse reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lai X, Cheng D, Xu H, Wang J, Lv X, Yao H, Li L, Wu J, Ye S, Li Z. Phase I Trial of Upamostat Combined With Gemcitabine in Locally Unresectable or Metastatic Pancreatic Cancer: Safety and Preliminary Efficacy Assessment. Cancer Med. 2025 Jan;14(1):e70550. doi: 10.1002/cam4.70550. PMID 39739976